CLINICAL TRIAL: NCT04806711
Title: Eleven Years of Menicon Z Night Contact Lens Wear in Reducing Myopia Progression in Children
Acronym: MCOS11
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menicon Co., Ltd. (Industry)
Collaborators: Universidad Europea de Madrid (Other); Clinica novovision (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCOS11
Record Dates: First submitted 2021-03-10; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Myopia, Progressive; Children, Only
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, parallel, longitudinal
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menicon Z Night (Experimental): The experimental arm consist of a group of Menicon Z Night orthokeratology contact lens wearers
  Interventions: Device: Menicon Z Night
- Control (Active Comparator): The active comparator arm consist of a control group of distance, single-vision glasses and contact lens wearers
  Interventions: Device: Control

INTERVENTIONS:
Device: Menicon Z Night — Menicon Z Night orthokeratology contact lenses were used to assess their efficacy in reducing myopia progression in children
  Arms: Menicon Z Night
Device: Control — Distance, single-vision glasses were used as a control
  Arms: Control

SUMMARY:
To compare axial length growth of white European myopic children wearing Menicon Z Night orthokeratology contact lenses to a control group of distance, single-vision glasses and contact lenses over an 11-year period.

DETAILED DESCRIPTION:
This prospective, controlled, parallel, longitudinal study compared the axial length growth of white European myopic children wearing Menicon Z Night orthokeratology contact lenses to a control group of distance, single-vision glasses and or distance, single-vision soft contact lenses over an 11-year period.

ELIGIBILITY:
Inclusion Criteria:

* Be 6 to 12 years of age, both ages inclusive
* A low-to-moderate level of myopia (between 0.75 and 4.00 D) and of astigmatism (≤ 1.00 D)
* Neophyte contact lens wearer
* Be successfully fitted with spectacles or orthokeratology contact lenses
* Be able to achieve, through spherical refraction correction, a logMAR visual acuity of 0.8 or better in each eye
* Be willing and able to follow the subject instructions and to meet the protocol-specified schedule of follow-up visits
* White European ethnicity

Exclusion Criteria:

* Systemic or ocular disease affecting ocular health
* Use of any systemic or topical medications that could affect ocular physiology or contact lens performance
* Any lid or anterior segment abnormalities for which contact lens wear could be contraindicated
* CCLRU grade ≥ 2 for any given anterior segment ocular clinical signs
* Aphakic, amblyopic, and atopic individuals
* Refractive astigmatism ≥ ½ spherical refraction
* Previous contact lens wear

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — White European
Enrollment: 20 (Actual)
Dates: Start 2007-03-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Axial length | 11 years
  To compare axial length growth of white European myopic children wearing Menicon Z Night orthokeratology contact lenses to a control group of distance, single-vision glasses and soft contact lens wearers. Measurements of axial length were taken with the Zeiss IOLMaster (Carl Zeiss Jena GmbH, Jena, Germany). Three separate measurements of axial length were recorded per subject and per visit, and a mean obtained.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Santodomingo-Rubido J, Villa-Collar C, Gilmartin B, Gutierrez-Ortega R. Myopia control with orthokeratology contact lenses in Spain: refractive and biometric changes. Invest Ophthalmol Vis Sci. 2012 Jul 31;53(8):5060-5. doi: 10.1167/iovs.11-8005. PMID 22729437
- [Result] Santodomingo-Rubido J, Villa-Collar C, Gilmartin B, Gutierrez-Ortega R, Sugimoto K. Long-term Efficacy of Orthokeratology Contact Lens Wear in Controlling the Progression of Childhood Myopia. Curr Eye Res. 2017 May;42(5):713-720. doi: 10.1080/02713683.2016.1221979. Epub 2016 Oct 21. PMID 27767354